CLINICAL TRIAL: NCT04590248
Title: A Phase 2b, Open-label, Single-arm, Multi-centre Study Assessing the Efficacy and Safety of Adavosertib as Treatment for Recurrent or Persistent Uterine Serous Carcinoma
Brief Title: A Study of Adavosertib as Treatment for Uterine Serous Carcinoma
Acronym: ADAGIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D601HC00002
Record Dates: First submitted 2020-09-22; First posted 2020-10-19 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Uterine Serous Carcinoma
Keywords: Adavosertib; Phase 2b; open-label; single-arm
MeSH Terms: interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adavosertib (Experimental): Subjects will receive adavosertib 300 mg administered orally, once daily on Days 1 to 5 and Days 8 to 12 of a 21-day treatment cycle.
  Interventions: Drug: Adavosertib

INTERVENTIONS:
Drug: Adavosertib — The subjects will receive oral adavosertib 300 mg, once daily on Days 1 to 5 and Days 8 to 12 of a 21-day treatment cycle.
  Other Names: AZD1775

SUMMARY:
This Phase 2b study aims to evaluate the efficacy and safety of adavosertib, an inhibitor of the tyrosine kinase WEE1, in subjects with recurrent or persistent uterine serous carcinoma (USC) who have previously received at least 1 prior platinum-based chemotherapy regimen for the management of USC.

DETAILED DESCRIPTION:
This Phase 2b, open-label, single-arm, multi-center study will assess the efficacy and safety of adavosertib in eligible subjects with histologically confirmed recurrent or persistent USC, evidence of measurable disease as per Response Evaluation Criteria in Solid Tumors.(RECIST) v1.1, and who have received at least 1 prior platinum-based chemotherapy regimen for the management of USC. Subjects with carcinosarcomas are not eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be aged ≥ 18 years of age inclusive, at the time of signing the informed consent.
2. Histologically confirmed recurrent or persistent USC. Subjects with carcinosarcomas are not eligible.
3. Evidence of measurable disease as per RECIST v1.1.
4. At least 1 prior platinum-based chemotherapy regimen for the management of USC. Prior receipt of immune checkpoint inhibitors, vascular endothelial growth factor (VEGF) inhibitors and human epidermal growth factor receptor 2 (HER2) targeted therapy is allowed. There is no restriction on the number of prior lines of systemic therapy.
5. Eastern Cooperative Oncology Group performance (ECOG) status 0-1.
6. Life expectancy ≥ 12 weeks.
7. Subjects must have normal organ and marrow function at baseline, within 7 days prior to study drug administration.
8. Consent to submit and provide a mandatory Formalin-fixed paraffin-embedded tumor sample for central testing.
9. Female subjects who are not of childbearing potential and women of childbearing potential who agree to use adequate contraceptive measures.

Exclusion Criteria:

1. Any underlying medical condition and uncontrolled intercurrent illness that would impair the ability of the subject to receive study treatment, as judged by the investigator.
2. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment.
3. Unable to swallow oral medications.
4. Spinal cord compression or metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study intervention.
5. Subjects with current signs or symptoms of bowel obstruction, including sub-occlusive disease, related to underlying disease.
6. Any of the following cardiac diseases currently or within the last 6 months:

   * Unstable angina pectoris
   * Acute myocardial infarction
   * Congestive heart failure
   * Conduction abnormality not controlled with pacemaker or medication
   * Significant ventricular or supraventricular arrhythmias
7. History of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected.
8. a) Resting corrected QTc interval using the Fridericia formula (QTcF) > 480 msec, or b) congenital long QT syndrome.
9. Immunocompromised subjects.
10. Subjects with known active hepatitis (ie, hepatitis B or C).
11. Prior treatment with any of the following:

    * Cell cycle checkpoint inhibitor.
    * Anticancer treatment drug ≤ 21 days (≤ 6 weeks for nitrosoureas or mitomycin C) or use of an investigational product within 5 half-lives prior to the first dose of adavosertib. For Programmed cell death-1 receptor (PD-1) /Programmed death-ligand 1 (PD-L1) inhibitors, a minimum of 28 days since last dose is required.
    * Prescription or non-prescription drugs known as moderate to strong inhibitors / inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment.
    * Herbal medications 7 days prior to first dose of study treatment.
12. Palliative radiotherapy with a limited field of radiation within 2 weeks or with wide field of radiation within 4 weeks prior to the first dose of study intervention.
13. Major surgical procedures ≤ 28 days, or minor surgical procedures ≤ 7 days, prior to beginning study.
14. Subjects with a known hypersensitivity or contraindication to adavosertib or any of the excipients of the product.
15. Currently pregnant or breast-feeding.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Liu, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (26):
- United States (14):
  - Research Site, Burbank, California
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, West Hollywood, California
  - Research Site, Aurora, Colorado
  - Research Site, Iowa City, Iowa
  - Research Site, Covington, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Spokane, Washington
  - Research Site, Vancouver, Washington
- Research Site, Toronto, Canada
- France (5):
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Herblain
- Italy (3):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
- Spain (3):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries and Associations Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Liu JF, Colombo N, Oza AM, Frenel JS, Corr BR, Rubinstein MM, Nevadunsky NS, Lheureux S, Gaba L, Gonzalez Cortijo L, Salutari V, You B, Chiang S, O'Connor MJ, Oplustil O'Connor L, Meulendijks D, Khatun M, Ghiorghiu D, Oaknin A. ADAGIO: A Phase IIb, Open-Label, Single-Arm, Multicenter Study Assessing the Efficacy and Safety of Adavosertib (AZD1775) as Treatment for Recurrent or Persistent Uterine Serous Carcinoma. J Clin Oncol. 2025 Sep 10;43(26):2897-2907. doi: 10.1200/JCO-24-01606. Epub 2025 Apr 22. PMID 40262070
- [Derived] Liu J, Oza AM, Colombo N, Oaknin A. ADAGIO: a phase IIb international study of the Wee1 inhibitor adavosertib in women with recurrent or persistent uterine serous carcinoma. Int J Gynecol Cancer. 2022 Jan;32(1):89-92. doi: 10.1136/ijgc-2021-003144. Epub 2021 Oct 29. PMID 34716177
- See also: D601HC00002_CSR_Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D601HC00002&attachmentIdentifier=2614291a-44ef-4b4b-a58a-844ac45c6899&fileName=D601HC00002_CSR_Synopsis_redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D601HC00002&attachmentIdentifier=1b089c0f-8c83-49cc-972c-f1fb195dcbe5&fileName=D601HC00002_SAP_redacted.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D601HC00002&attachmentIdentifier=3e63fd57-34c2-4bbc-a694-bf7eabd353ea&fileName=D601HC00002_CSP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 sites in 5 countries (United States, Canada, France, Italy and Spain) from 30-November-2020 to 07-February-2023.
Pre-assignment Details: Participants had been through a screening period of 28 days, followed by assessments as per schedule of activities.
Groups:
- Adavosertib: Participants received adavosertib 300 mg administered orally, once daily on Days 1 to 5 followed by 2 days off and Days 8 to 12 (21 days treatment cycle).
Period: Overall Study
Arm/Group | Adavosertib
Started | 109
Completed | 90
Not Completed | 19
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 16
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Full-analysis set (FAS), which included all participants who received at least one (non-zero) dose of study treatment.
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African or American | 9
  Asian | 1
  White | 92
  Other | 3
  Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 for target lesions (TLs) and assessed by computed tomography (CT) or magnetic resonance imaging (MRI): Complete response (CR), Disappearance of all target lesions; Partial response (PR), >=30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: up to 75 weeks
Population: FAS, which included all participants who received at least one (non-zero) dose of study treatment. Here, overall number of participants analyzed signifies the participant with available data that were analyzed for the outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adavosertib
Number analyzed (Participants) | 104
Percentage of participants | 26 [17.9 to 35.5]

2. Secondary Outcome: Duration of Response (DoR)
Description: The time from the date of first documented response until date of documented progression per RECIST v1.1 as assessed by BICR, or death in the absence of disease progression
Time Frame: up to 75 weeks
Population: FAS, which included all participants who received at least one (non-zero) dose of study treatment and had a confirmed response.
Measure: Median (Full Range); unit: Months
Arm/Group | Adavosertib
Number analyzed (Participants) | 27
Months | 4.7 [1.4 to 10.5]

3. Secondary Outcome: Depth of Response
Description: Depth of response is defined as best percentage change from baseline in target lesion size, which is the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction. A negative change denotes a reduction in target lesion size.
Time Frame: Up to 75 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Adavosertib
Number analyzed (Participants) | 100
Percentage change | -20.8 (31.60)

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from first dose until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraws from study drug or receives another anticancer therapy prior to progression. PFS was assessed per RECIST v1.1 using CT or MRI scans by BICR.
Time Frame: Up to 75 weeks
Population: FAS, which included all participants who received at least one (non-zero) dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
Months | 2.8 [2.60 to 3.94]

5. Secondary Outcome: Progression Free Survival Rate at 6 Months (PFS6)
Description: The progression free survival rate was assessed at 6 months by Kaplan-Meier estimate per RECIST v1.1.
Time Frame: Up to 6 months
Population: FAS, which included all participants who received at least one (non-zero) dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
Percentage | 18.1 [10.42 to 27.55]

6. Secondary Outcome: Overall Survival (OS)
Description: The time from date of first dose until the date of death due to any cause
Time Frame: Up to 75 weeks
Population: FAS, which included all participants who received at least one (non-zero) dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
Months | 9.6 [8.28 to NA] — Not calculable due to lack of events near the median.

7. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of participants who have a best overall response of confirmed response (CR) or partial response (PR) or who have stable disease for at least 5 weeks after start of treatment, based on BICR.
Time Frame: Up to 75 weeks
Population: FAS, which included all subjects who received at least one (non-zero) dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
Percentage of participants | 51.4 [41.6 to 61.1]

8. Secondary Outcome: Lowest Concentration (Ctrough) of Adavosertib
Description: Lowest plasma concentration of adavosertib was evaluated as pharmacokinetic paramerter.
Time Frame: Cycle 1, Day 5 and Cycle 2, Day 5 (pre-dose) (each cycle is 21 days)
Population: The pharmacokinetic analysis set included all dosed participants who had at least one measurable plasma concentration collected post-dose which was obtained without any deviation or event thought to significantly affect the pharmacokinetic analysis. Here, overall number of participants analyzed signifies in each row the participant with available data, that was analyzed for specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nM)
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
nanomole (nM)
  Cycle 1 Day 5: number analyzed (Participants) | 91
  Cycle 1 Day 5 | 307.2 (105.6)
  Cycle 2 Day 5: number analyzed (Participants) | 79
  Cycle 2 Day 5 | 328.7 (70.3)

9. Secondary Outcome: Maximum Concentration (Cmax) of Adavosertib
Description: Maximum plasma concentration of adavosertib was evaluated as pharmacokinetic parameter.
Time Frame: Cycle 1, Day 5 and Cycle 2, Day 5 (2 hours post-dose) (each cycle is 21 days)
Population: The pharmacokinetic analysis set included all dosed participants who had at least one measurable plasma concentration collected post-dose which was obtained without any deviation or event thought to significantly affect the pharmacokinetic analysis. Here, overall number of participants analyzed in each row signifies the participant with available data, that was analyzed for specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
nM
  Cycle 1 Day 5: number analyzed (Participants) | 83
  Cycle 1 Day 5 | 1115.9 (82.1)
  Cycle 2 Day 5: number analyzed (Participants) | 72
  Cycle 2 Day 5 | 1356.5 (59.3)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: The number of participants with treatment emergent adverse events (AEs) were assessed as variable of safety and tolerability. The adverse events reported here were treatment emergent.
Time Frame: From baseline to post-treatment follow-up (30 days after last dose), approximately up to 114 weeks
Population: FAS, which included all participants who received at least one (non-zero) dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Adavosertib
Number analyzed (Participants) | 109
Participants
  Any AE | 109
  Any AE possibly related to treatment | 106
  Any AE with outcome = death | 4
  Any AE with outcome = death, possibly related to treatment | 1
  Any AE of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher | 75
  Any AE of CTCAE grade 3 or higher, possibly related to treatment | 66
  Any AE leading to discontinuation of IP | 19
  Any AE leading to discontinuation of IP, possibly related to treatment | 16
  Any serious adverse event (SAE) (including events with outcome = death) | 50
  Any SAE (including events with outcome = death), possibly related to treatment | 29
  Any SAE leading to discontinuation of investigational product (IP) | 10
  Any SAE leading to discontinuation of IP, possibly related to treatment | 8
  Any AE leading to dose modification of IP | 79
  Any AE leading to dose reduction of IP | 62
  Any AE leading to dose interruption of IP | 72
  Any AE leading to dose interruption possibly related to treatment | 62
  Any AE leading to dose reduction possibly related to treatment | 60

ADVERSE EVENTS:
Time Frame: From baseline to post-treatment follow-up (30 days after last dose), approximately up to 114 weeks
Description: All adverse events during the trial are reported.
Arm/Group | Adavosertib
All-Cause Mortality (participants affected / at risk) | 47/109
Serious Adverse Events (participants affected / at risk) | 53/109
Other Adverse Events (participants affected / at risk) | 109/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adavosertib (N=109)
Biliary sepsis (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Embolism (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adavosertib (N=109)
Urinary tract infection (Infections and infestations) | 16 (19)
Anaemia (Blood and lymphatic system disorders) | 74 (155)
Leukopenia (Blood and lymphatic system disorders) | 8 (15)
Neutropenia (Blood and lymphatic system disorders) | 26 (48)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (40)
Decreased appetite (Metabolism and nutrition disorders) | 27 (39)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (21)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (27)
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 (27)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (11)
Insomnia (Psychiatric disorders) | 9 (9)
Dizziness (Nervous system disorders) | 11 (17)
Dysgeusia (Nervous system disorders) | 17 (19)
Headache (Nervous system disorders) | 14 (19)
Hypertension (Vascular disorders) | 15 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (21)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 34 (45)
Abdominal pain upper (Gastrointestinal disorders) | 16 (22)
Constipation (Gastrointestinal disorders) | 45 (58)
Diarrhoea (Gastrointestinal disorders) | 73 (146)
Dyspepsia (Gastrointestinal disorders) | 13 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 71 (140)
Vomiting (Gastrointestinal disorders) | 39 (55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Dysuria (Renal and urinary disorders) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 7 (7)
Asthenia (General disorders) | 45 (72)
Fatigue (General disorders) | 43 (66)
Non-cardiac chest pain (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 20 (26)
Pyrexia (General disorders) | 7 (8)
Alanine aminotransferase increased (Investigations) | 28 (39)
Aspartate aminotransferase increased (Investigations) | 23 (31)
Blood alkaline phosphatase increased (Investigations) | 14 (18)
Blood creatinine increased (Investigations) | 27 (40)
Lymphocyte count decreased (Investigations) | 6 (9)
Neutrophil count decreased (Investigations) | 16 (31)
Platelet count decreased (Investigations) | 22 (40)
Weight decreased (Investigations) | 12 (16)
Fall (Injury, poisoning and procedural complications) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT04590248/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT04590248/SAP_001.pdf